CLINICAL TRIAL: NCT03985735
Title: Characterisation of Gut Microbiota, Bispectral Index Data and Plasma Kynurenine in Patients Undergoing Video-assisted Thoracic Surgery
Status: Completed | Type: Observational
Sponsor: China Medical University, China (Other)
Responsible Party: Principal Investigator, Wen-fei Tan, Professor, China Medical University, China
Other Study IDs: 20190609
Record Dates: First submitted 2019-06-07; First posted 2019-06-14 (Actual); Last update posted 2020-06-22 (Actual); Status verified 2020-06

CONDITIONS: Lung Cancer
MeSH Terms: conditions — Lung Neoplasms | interventions — Anesthesia, General

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Group good sleepers: Duration of sleep was defined as the duration of all Bispectral Index data below 80 in the 12 hours of monitoring (from 20:00pm to 06:00am).
  Sleeping time are more than six hours.
  Interventions: Drug: General anesthesia
- Group poor sleepers: Duration of sleep was defined as the duration of all Bispectral Index data below 80 in the 12 hours of monitoring (from 20:00pm to 06:00am).
  Sleeping time are less than two hours.
  Interventions: Drug: General anesthesia

INTERVENTIONS:
Drug: General anesthesia — For maintenance of propofol anesthesia, total intravenous anesthesia was administered by using propofol (Fresenius Kabi, Austria GmbH) at a plasma target concentration (Marsh pharmacokinetic model software) of 2.5-4 μg/ml. Remifentanil (0.2-0.5 μg/kg/min) was given to all patients during the operation. Additional cisatracurium （0.05 mg/kg）and fentanyl (30-50 μg at the end of surgery) were used as needed, in accordance with the clinical requirements.

SUMMARY:
The study is a case-controlled observational trial. Sixty patients will be divided into 2 groups (good or poor sleepers) depending on their first postoperative night Bispectral index data. Firstly, this study aims to characterise the gut and lung microbiota in patients with lung cancer treated with surgery. Secondly, it aims to evaluate microbiota and its influence on plasma kynurenine.

DETAILED DESCRIPTION:
The study is a case-controlled observational trial. Sixty patients will be divided into 2 groups (good or poor sleepers) depending on their first postoperative night Bispectral index data. Firstly, this study aims to characterise the gut and lung microbiota in patients with lung cancer treated with surgery. Secondly, it aims to evaluate microbiota and its influence on plasma kynurenine.

ELIGIBILITY:
Inclusion Criteria:

* 1. ethnic Chinese;
* 2. age, 18 to 75 years old;
* 3. American Society of Anaesthesiologists (ASA) physical status I or II;
* 4. required VATS for lung surgery and one lung ventilation .

Exclusion Criteria:

* Cognitive difficulties
* Partial or complete gastrectomy
* Previous esophageal surgery
* Previous treated by radiotherapy or surgery
* Inability to conform to the study's requirements
* body mass index exceeding 30 kg/m2
* Deprivation of a right to decide by an administrative or juridical entity
* Ongoing participation or participation in another study <1 month ago
* preoperative Pittsburgh Sleep Quality Index global scores higher than 6
* recent (< 3 months prior) use of antibiotics, probiotics, prebiotics, symbiotics, hormonal medication, laxatives, proton pump inhibitors, insulin sensitizers or traditional Chinese medicine

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Gender Based: Yes — male
Study Population: The study is a case-controlled observational trial. Sixty patients will be divided into 2 groups (good or poor sleepers) depending on their first postoperative night Bispectral index data.
Sampling Method: Non-Probability Sample
Enrollment: 20 (Actual)
Dates: Start 2019-08-01 (Actual); Primary Completion 2019-12-31 (Actual); Study Completion 2020-01-20 (Actual)

PRIMARY OUTCOMES:
lung and gut microbiota | from baseline to postoperative 72 hours
  this study will characterise the lung and gut microbiota in 2 groups of 30 patients

SECONDARY OUTCOMES:
Bispectral index data | the first postoperative night
  this study will characterise the Bispectral index data in 2 groups of 30 patients
plasma kynurenine concentrations | baseline and the first postoperative night
  this study will characterise the plasma kynurenine concentrations in 2 groups of 30 patients

CONTACTS AND LOCATIONS:
Locations (1):
- the First Hospital of China Medical University, Shenyang, Liaoning, China